CLINICAL TRIAL: NCT00080613
Title: Phase II Study of Neoadjuvant and Adjuvant Exemestane in Postmenopausal Women With Locally Advanced Hormone Receptor-Positive Breast Cancer
Brief Title: Neoadjuvant and Adjuvant Exemestane in Treating Postmenopausal Women With Locally Advanced Hormone Receptor-Positive Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Robert H. Lurie Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU-02B4; CDR0000346457 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Chemotherapy, Adjuvant; Aromatase Inhibitors; Neoadjuvant Therapy; Surgical Procedures, Operative

INTERVENTIONS:
Drug: exemestane
Procedure: adjuvant therapy
Procedure: aromatase inhibition
Procedure: conventional surgery
Procedure: endocrine therapy
Procedure: hormone therapy
Procedure: neoadjuvant therapy
Procedure: surgery

SUMMARY:
RATIONALE: Estrogen and progesterone can stimulate the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by reducing the production of estrogen and progesterone. Giving hormone therapy before surgery may shrink the tumor so it can be removed with breast-conserving surgery. Giving hormone therapy after surgery may kill any remaining tumor cells.

PURPOSE: Phase II trial to study the effectiveness of neoadjuvant and adjuvant exemestane in treating postmenopausal women who have locally advancedestrogen and/or progesterone receptor-positive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in postmenopausal women with locally advanced hormone receptor-positive breast cancer treated with neoadjuvant and adjuvant exemestane.

Secondary

* Determine the response rate by mammography, ultrasound, MRI, and positron emission tomography scan in patients treated with this drug.
* Determine the time to progression in patients treated with this drug.
* Compare the expression of hormone receptors and epidermal growth factor receptors (including HER2/neu) in patients prior to and after treatment with this drug and correlate these results with clinical response rates.

OUTLINE: Patients receive oral exemestane once daily for 16 weeks in the absence of disease progression or unacceptable toxicity. After 16 weeks, patients undergo surgery and then continue exemestane once daily for a total of 5 years (including the 16 weeks before surgery).

Patients are followed every 3 months for 2 years after surgery and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 16-46 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer
* Locally advanced disease (stage II or III)
* Not amenable to breast-conserving therapy at the time of diagnosis
* Measurable disease meeting 1 of the following criteria:
* Bidimensionally measurable palpable lesion at least 1 cm by caliper
* Unidimensionally measurable lesion at least 1 cm by a positive mammogram, ultrasound, or MRI
* No evidence of disease outside the breast or chest wall except ipsilateral axillary lymph nodes
* Hormone receptor status:
* Estrogen and/or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, defined as any of the following:
* Over 60 years of age
* Over 45 years of age with an intact uterus and amenorrhea for more than 12 months
* Prior hysterectomy with follicle-stimulating hormone levels within the postmenopausal range
* Prior ovarian ablation (i.e., bilateral surgical)

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)

Renal

* Creatinine less than 2 mg/dL

Other

* No other prior or concurrent cancer except nonmetastatic nonmelanoma skin cancer, carcinoma in situ of the cervix, or cancer cured by surgery within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for breast cancer

Chemotherapy

* No prior chemotherapy for breast cancer

Endocrine therapy

* No prior hormonal therapy for breast cancer

Radiotherapy

* No prior radiotherapy for breast cancer

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William John Gradishar, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States